CLINICAL TRIAL: NCT05597137
Title: To Explore the Regulatory Effect of Zinc on Intestinal Flora in Healthy Adults # A Single-center, Prospective, Self-controlled Trial
Brief Title: The Exploration of the Regulatory Effect of Zinc on Intestinal Flora in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Seventh Affiliated Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Yu Chen, chief physician, The Seventh Affiliated Hospital, Southern Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: (2022)--0008
Record Dates: First submitted 2022-10-24; First posted 2022-10-27 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Healthy
Keywords: Zinc, gut microbiota, healthy adult
MeSH Terms: interventions — gluconic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): During the study period, all subjects were required to avoid a diet high in zinc in order to avoid interference with dietary zinc intake and reduce bias in the weeks 1-2. In the weeks 3-4, all subjects were started to receive zinc supplementation at the normal adult dose (zinc tablets: 1 tablet (10mg Zinc) once daily after meals), while maintaining the avoidance of high-zinc foods.
  Interventions: Dietary Supplement: Zinc Gluconate

INTERVENTIONS:
Dietary Supplement: Zinc Gluconate — Each participant should receive a regular zinc diet for weeks 1-2 and take zinc supplements for weeks 3-4.

SUMMARY:
In this A Single-center, Prospective, Self-controlled trial, subjects should avoid a high-Zinc diet for 2 weeks and then take Zinc supplements for 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 20-30 years from the general community were recruited to participate in the study voluntarily without underlying diseases.

Exclusion Criteria:

Patients who have taken antibiotics orally in the past 3 months or have acute or chronic inflammation; Those who have taken hormones within 3 months; Have taken any drugs that may interfere with glucose and lipid metabolism (such as insulin, glyburide, indomethacin, phentolamine, fuuside, phenytoin sodium, cortisone, etc.) and have had probiotic intervention within 1 month; smokers and drinkers; Uncontrollable mental disorders (including hospitalization history of mental illness); (6) Currently attending a weight loss or weight management course; prescribed diet for specific or other reasons (e.g. celiac disease); pregnant or lactating women; Patients with cardiac and renal insufficiency; Patients with other underlying diseases; Long-term constipation.

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
16S rDNA sequencing | 14days，28 days
  16S rDNA sequencing technology was used to identify the structural and functional changes of intestinal microbiota before and after Zinc supplementation.
metabolomic analysis of serum and feces | 14days，28 days
  To determine the alteration of gut microbiota after Zn supplementary.
The blood levels of Zn2+ in each study phase | 14days，28 days
  The blood levels of Zn2+ would be detected on day 14 and day 28.
Number of participantswith abnormal laboratory tests results | 14days，28 days
  If there are abnormal situations during the experiment that may pose significant risks to the health or safety of the participants, the research team may need to terminate the experiment to ensure participant safety. Only
The fecal Zn2+ concentration in each study phase | 14days，28 days
  The fecal Zn2+ concentration would be detected on day 14 and day 28.

SECONDARY OUTCOMES:
Total bilirubin concentration after 14days oral Zn. | 14days，28 days
  change from 14days in Total bilirubin and analyzed by the AU5800 fully automatic biochemical analyzer.
Direct bilirubin concentration after 14days oral Zn. | 14days，28 days
  change from 14days in Direct bilirubin and analyzed by the AU5800 fully automatic biochemical analyzer.
Indirect bilirubin concentration after 14days oral Zn. | 14days，28 days
  change from 14days in indirect bilirubin and analyzed by the AU5800 fully automatic biochemical analyzer.
uric acid concentration after 14days oral Zn. | 14days，28 days
  change from 14days in uric acid and analyzed by the AU5800 fully automatic biochemical analyzer.
total triglyceride concentration after 14days oral Zn. | 14days，28 days
  change from 14days in total triglyceride and analyzed by the AU5800 fully automatic biochemical analyzer.
total protein concentration after 14days oral Zn. | 14days，28 days
  change from 14days in total protein and analyzed by the AU5800 fully automatic biochemical analyzer.
aspartate transaminase concentration after 14days oral Zn. | 14days，28 days
  change from 14days in aspartate transaminase and analyzed by the AU5800 fully automatic biochemical analyzer.
alanine transaminase concentration after 14days oral Zn. | 14days，28 days
  change from 14days in alanine transaminase and analyzed by the AU5800 fully automatic biochemical analyzer.
albumin concentration after 14days oral Zn. | 14days，28 days
  change from 14days in albumin and analyzed by the AU5800 fully automatic biochemical analyzer.
total cholesterol concentration after 14days oral Zn. | 14days，28 days
  change from 14days in total cholesterol and analyzed by the AU5800 fully automatic biochemical analyzer.
Urea concentration after 14days oral Zn. | 14days，28 days
  change from 14 days in urea and analyzed by the AU5800 fully automatic biochemical analyzer.
HDL-C concentration after 14days oral Zn. | 14days，28 days
  change from 14 days in HDL-C(high density lipoprotein cholesterol) and analyzed by the AU5800 fully automatic
LDL-C concentration after 14days oral Zn. | 14days，28 days
  change from 14 days in LDC-C(low density lipoprotein cholesterol) and analyzed by the AU5800 fully automatic
Red blood cells analysis after 14days oral Zn. | 14days，28 days
  change from 14days in Red blood cells and determined by a Sysmex-xn-2000 automatic blood cell analyser.
Plateltes analysis after 14days oral Zn. | 14days，28 days
  change from 14 days in Plateltes and determined by a Sysmex-xn-2000 automatic blood cell analyser.
Neutrophil cells analysis after 14days oral Zn. | 14days，28 days
  change from 14days in Neutrophil cells and determined by a Sysmex-xn-2000 automatic blood cell analyser.
Eosinophil cells analysis after 14days oral Zn. | 14days，28 days
  change from 14days in Eosinophil cells and determined by a Sysmex-xn-2000 automatic blood cell analyser.
Basophil cells analysis after 14days oral Zn. | 14days，28 days
  change from 14 days in Basophil cells and determined by a Sysmex-xn-2000 automatic blood cell analyser.
Lymphocyte cells analysis after 14days oral Zn. | 14days，28 days
  change from 14 days in Lymphocyte cells and determined by a Sysmex-xn-2000 automatic blood cell analyser.
Monocyte cells analysis after 14days oral Zn. | 14days，28 days
  change from 14 days in Monocyte cells and determined by a Sysmex-xn-2000 automatic blood cell analyser.
White blood cells analysis after 14days oral Zn. | 14days，28 days
  change from 14 days in white blood cells and determined by a Sysmex-xn-2000 automatic blood cell analyser.

CONTACTS AND LOCATIONS:
Locations (1):
- Southern Medical Unversity，the seventh affiliated hospital, Foshan, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Since some data may involve subject's privacy #we have no plans to share data so far# and some data may be shared later depending on the subjects's wishes.

REFERENCES:
- [Background] Ackland ML, Michalczyk AA. Zinc and infant nutrition. Arch Biochem Biophys. 2016 Dec 1;611:51-57. doi: 10.1016/j.abb.2016.06.011. Epub 2016 Jun 15. PMID 27317042
- [Derived] Li D, Wan M, Xue L, Zhang Z, Qiu Y, Mei F, Tang N, Yu C, Yu Y, Chen T, Ding X, Yang Q, Liu Q, Gu P, Jia W, Chen Y, Chen P. Zinc promotes microbial p-coumaric acid production that protects against cholestatic liver injury. Cell Host Microbe. 2024 Dec 11;32(12):2195-2211.e9. doi: 10.1016/j.chom.2024.11.002. Epub 2024 Nov 27. PMID 39610253
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/27317042/